CLINICAL TRIAL: NCT04555109
Title: Convalescent Plasma for COVID-19 Research (CONCOR) Donor Study
Brief Title: Convalescent Plasma for COVID-19 Research Donor Study
Acronym: CONCOR-Donor
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Rulan Parekh, Staff Physician, Associate Chief Clinical Research, The Hospital for Sick Children
Other Study IDs: 1000070462
Record Dates: First submitted 2020-09-17; First posted 2020-09-18 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Covid19
Keywords: Covid19; Convalescent plasma; Seroconversion; Immunity; National; Biorepository; Observational Study
MeSH Terms: conditions — COVID-19; HIV Seropositivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Specimen collection will include DNA, serum, plasma, peripheral blood mononuclear cells and whole blood.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID-19 Convalescents: The cohort will include up to 1000 persons recovered from COVID-19, ages 17 - 65, that will provide a written consent form to participate in the study, complete questionnaires and provide a blood sample.

SUMMARY:
Convalescent Plasma for COVID-19 Research (CONCOR-Donor) study, is a national, natural history study of plasma donors recovered from COVID-19. CONCOR-Donor study will address immune response, duration of protective immunity, and clinical factors and host genetics contributing to the variability of immune response. We will also study long-term outcomes from COVID-19 infection. Results from the study will help define therapeutic strategies for COVID-19.

DETAILED DESCRIPTION:
The outbreak caused by Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) led to the global pandemic. There are currently no proven treatments for coronavirus disease (COVID-19), however, convalescent plasma has emerged as a potential therapeutic to prevent clinical deterioration. Convalescent plasma was successfully used for other infections, in small numbers, but there is limited evidence for the efficacy of administering specific, neutralizing antibodies by transfusion of convalescent plasma. The unknown role for convalescent plasma in treating COVID-19 necessitates further study.

As trials are underway to determine efficacy of using convalescent plasma, we will use this unique opportunity to conduct a national longitudinal cohort study of 1000 persons recovered from COVID-19 and volunteer to donate convalescent plasma. Our aims are to:1) determine if the variability of titers of viral neutralizing antibody and ELISA antibody are associated with clinical and demographic factors; 2) determine duration of protective immunity in recovered persons over 1 year and if modified by clinical and demographic factors; 3) determine genetic risk predictors of the antibody response, and 4) create a biorepository available to researchers from across Canada. Based on the World Health Organization (WHO) Coordinated Global Research Map, this project addresses the priority of the natural history of COVID-19 and clinical characterization of antibody response in the convalescent phase and beyond.

ELIGIBILITY:
Inclusion Criteria:

* Recovered from COVID-19 infection
* Have a positive PCR or serology or a positive household contact
* Signed informed consent form
* Provide blood sample
* Ability to complete a questionnaire

Exclusion Criteria:

* None

Ages: 17 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All that recovered from COVID-19 above age 17, that have tested positive or a household contact that tested positive regardless of eligibility to donate plasma for the trials.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2020-06-30 (Actual); Primary Completion 2022-10-30 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
Seroprevalence and duration of protective immunity | 12 months
  Determine if the titers of SARS-CoV-2-specific neutralizing antibody and serum ELISA antibodies, are correlated with clinical and demographic factors such as age, sex, comorbidities, geographic region, and severity of prior COVID-19 symptoms, during the convalescent phase.

CONTACTS AND LOCATIONS:
Overall Officials: Rulan Parekh, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No